CLINICAL TRIAL: NCT06061003
Title: Can High Resolution 3D Resin Printed Models be Used in Clinical Anatomy Education for Fracture Rehabilitation
Brief Title: 3D Resin Printed Fracture Models for Anatomy Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assist. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-FTR-RK-08
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Educational Problems; Anatomical Pathological Condition
MeSH Terms: conditions — Pathological Conditions, Anatomical

STUDY DESIGN:
Intervention Model Description: Two groups as intervention and control groups. Assessments will be performed before intervention, and after the theorical/practical lectures.
Who Masked: Outcomes Assessor
Masking Description: Due to the study design, control group will not receive any fractured models for practical lectures therefore only outcome assessor will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractured Model Group (Other): All participants will receive 60 minutes training on anatomy and pathophysiology of theoric wrist fractures. After lecture completed, the Fractured Model Group will engage in a 2-hours hands-on practical session in the laboratory, working with wrist fracture models.
  Interventions: Other: Clinical Anatomical Education with Fractured Bone Models
- Standard Anatomic Model Group (Other): All participants will receive 60 minutes training on anatomy and pathophysiology of theoric wrist fractures.After lecture completed, the Standard Anatomic Model Group will engage in a 2-hours hands-on practical session in the laboratory, working with standard anatomical wrist models.
  Interventions: Other: Clinical Anatomical Education with Standard Bone Models

INTERVENTIONS:
Other: Clinical Anatomical Education with Fractured Bone Models — Participants will undergo a 2-hour training session, consisting of 60 minutes of theory and 60 minutes of practice. The theoretical lesson, supported by 2D images illustrating wrist anatomy, types of fractures, and rehabilitation based on fracture type, will be simultaneously delivered to both groups. Following this, the practical group will receive a 60-minute hands-on session using 3D-printed digital models of radius and ulna fractures. These training sessions will be scheduled in the morning hours, on a day when students have no other classes between 9 am and 12 pm, to minimize mental fatigue and exhaustion. In the practical session, anatomical structures, their relationships, and arrangements will be demonstrated to the practice group using a model of a fractured wrist.
  Arms: Fractured Model Group
Other: Clinical Anatomical Education with Standard Bone Models — Participants will undergo a 2-hour training session, consisting of 60 minutes of theory and 60 minutes of practice. The theoretical lesson, supported by 2D images illustrating wrist anatomy, types of fractures, and rehabilitation based on fracture type, will be simultaneously delivered to both groups. Following this, the practical group will receive a 60-minute hands-on session using 3D-printed digital models of radius and ulna fractures. These training sessions will be scheduled in the morning hours, on a day when students have no other classes between 9 am and 12 pm, to minimize mental fatigue and exhaustion. The control group will receive the same practical session using a standard anatomical model.
  Arms: Standard Anatomic Model Group

SUMMARY:
Resin printing is an emerging technology with a wide array of applications. This research seeks to assess the practicality of incorporating 3D resin printed models into anatomy education while investigating how fractured models impact students' decision-making and quiz scores.

DETAILED DESCRIPTION:
Over the past decade, 3D printing has become increasingly accessible and cost-effective, offering systems and materials suitable for home use. 3D printing is a technology that streamlines production by translating computer-generated models into physical objects, layer by layer. In comparison to other tissue engineering and rapid prototyping methods, 3D printing boasts numerous advantages, such as exceptional precision, rapid production, cost-effectiveness, and seamless integration. Utilizing 3D models can significantly enhance the comprehension of intricate structures for medical professionals and students alike. Common materials used in 3D printing include robust nylon, aluminum, gypsum, textile components, polylactic acid, and resin. Among these, photosensitive resin stands out, as it enables the creation of higher-quality, more intricate structures that closely resemble real tissues, offering a smoother finish devoid of visible raw material textures.

This study's primary objective was to assess the suitability of tissues produced by a 3D resin printer in anatomy education, with the aim of enhancing hands-on training through direct manipulation of fractured bone models.

ELIGIBILITY:
Inclusion Criteria:

* having stereopsis above 40 arc/seconds according to the Titmus Stereopsis Test

Exclusion Criteria:

* having partial or total vision loss
* having a history of traumatic injury to the upper extremities within the last six months
* having used wrist anatomy models in virtual or real environments

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Test | one hour
  A 25-question multiple choice questions test will be employed to assess students' anatomical knowledge and their decision-making capabilities for the rehabilitation program. The test will be prepared according to Bloom's taxonomy and will consist of both multiple-choice and open-ended questions. Total test time wil lbe 60 minutes and scores will be recorded as percentages.

SECONDARY OUTCOMES:
Academic Motivation | one hour
  Academic Motivation Scale test taking motivation questionnaire will be used to assess participants' motivations. This scale, consisting of 22 questions and 7 subscales, evaluates amotivation, as well as internal and external motivation.
Test Anxiety Inventory | one hour
  To examine whether there is a change in the level of anxiety experienced by students during the exam, a 5-question short version of Test Anxiety Inventory will be used. The test includes sections related to ease, comfort associated with learning, and alignment of exam questions with the course.
Enjoyment and Ease of Use Assessment | one hour
  Participants will fill out a feedback questionnaire regarding the learning instruments using visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Kurul, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kurul R, Inal B, Diramali M, Ozer H, Erdogan KE. Evaluating the educational impact of tomography-based high-resolution 3D-printed distal radius fracture models. BMC Med Educ. 2025 Dec 24;25(1):1706. doi: 10.1186/s12909-025-08164-w. PMID 41444874